CLINICAL TRIAL: NCT00661947
Title: Pharmacokinetics and Pharmacodynamics of Fructose Following Soft Drink Consumption: Sucrose vs High Fructose Corn Syrup
Brief Title: Pharmacokinetics and Pharmacodynamics of Fructose
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 682-2007
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: fructose; sucrose; high fructose corn syrup; serum uric acid; lactate; glucose; triglycerides; Bioavailability of fructose from two formulations
MeSH Terms: interventions — Sucrose; High Fructose Corn Syrup

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, whole blood, serum, plasma, and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Public: General public. Those who are not currently taking any medication besides birth control pills.
  Interventions: Other: Dr Pepper sweetened with sucrose or high fructose corn syrup

INTERVENTIONS:
Other: Dr Pepper sweetened with sucrose or high fructose corn syrup — Comparison of different formulations of fructose.

SUMMARY:
The purpose of this study is to determine whether sucrose vs high fructose corn syrup from a soft drink results in differences in various metabolic byproducts such as fructose, glucose, serum uric acid, triglyceride and lactate.

DETAILED DESCRIPTION:
Fructose consumption has risen sharply during the past several decades. Since its introduction to the United States in 1967, high fructose corn syrup (HFCS) has overtaken sucrose as the main sweetener in manufactured foods and beverages, and thus, is responsible for the approximately 30% increase in fructose in our diet. Numerous studies have shown that excessive fructose consumption can cause a variety of harmful metabolic effects, suggesting that fructose may partially be responsible for the current epidemic in obesity, hypertension, metabolic syndrome, and diabetes.

This preliminary study will investigate the pharmacokinetics and pharmacodynamics of fructose in a broad population. Specifically, the goal of our research are to compare the impact of the two main sources of dietary fructose, sucrose versus HFCS, on fructose bioavailability and acute metabolic changes by measuring response phenotypes, such as serum uric acid, lactate, and triglyceride levels.

ELIGIBILITY:
Inclusion Criteria:

* adult subjects aged 18 years or older
* either gender
* any ethnicity
* willing to abstain from drinking any alcohol 3 days prior to a study visit

Exclusion Criteria:

* history of liver or kidney disease
* history of diabetes mellitus or fasting blood glucose ≥ 126 mg/dl or random blood glucose ≥ 200 mg/dl
* currently taking any medication (except oral contraceptives)
* consume more than 1 alcoholic drink per day
* pregnant or breast-feeding
* blood donor in the previous 8 weeks
* history of gout

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population from Gainesville, FL area.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Fructose | baseline, 15min, 30 min, 60 min, 90 min, 2 hr, 3 hr, 4.5 hr, 6 hr

SECONDARY OUTCOMES:
serum uric acid | baseline, 15 min, 30 min, 60 min, 90 min, 2 hr, 3 hr, 4.5 hr, 6 hr
glucose | baseline, 15 min, 30 min, 60 min, 90 min, 2 hr, 3 hr, 4.5 hr, 6 hr
lactate | baseline, 15 min, 30 min, 60 min, 90 min, 2 hr, 3 hr, 4.5 hr, 6 hr
triglycerides | baseline, 15 min, 30 min, 60 min, 90 min, 2 hr, 3 hr, 4.5 hr, 6 hr

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Johnson, Pharm.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Department of Pharmacy Practice, Center for Pharmacogenomics, Gainesville, Florida, United States

REFERENCES:
- [Result] Le MT, Frye RF, Rivard CJ, Cheng J, McFann KK, Segal MS, Johnson RJ, Johnson JA. Effects of high-fructose corn syrup and sucrose on the pharmacokinetics of fructose and acute metabolic and hemodynamic responses in healthy subjects. Metabolism. 2012 May;61(5):641-51. doi: 10.1016/j.metabol.2011.09.013. Epub 2011 Dec 5. PMID 22152650